CLINICAL TRIAL: NCT04882124
Title: A 12-week Randomized, participant-and Investigator-blinded, Placebo-controlled, Parallel Group Study to Explore the Efficacy, Pharmacodynamics, Safety, and Pharmacokinetics of Two Doses of Inhaled CSJ117 in Adults With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Study of Effect of CSJ117 on Symptoms, Pharmacodynamics and Safety in Patients With COPD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCSJ117B12201
Record Dates: First submitted 2021-04-28; First posted 2021-05-11 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Chronic Obstructive Pulmonary Disease; COPD; CSJ117
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- CSJ117 8mg (Experimental): Intervention: Drug: CSJ117
  Interventions: Drug: CSJ117
- CSJ117 4mg (Experimental): Intervention: Drug: CSJ117
  Interventions: Drug: CSJ117
- CSJ117 Placebo (Placebo Comparator): Intervention: Drug: Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CSJ117 — CSJ117 (4 mg and 8 mg) inhaled once daily for 12 weeks. Delivered via Concept1 device.
  Arms: CSJ117 4mg; CSJ117 8mg
Drug: Placebo — Placebo inhaled once daily for 12 weeks. Delivered via Concept1 device
  Arms: CSJ117 Placebo

SUMMARY:
This is a Phase 2 study in patients with chronic obstructive pulmonary disease (COPD) to assess the efficacy, pharmacodynamics (PD), pharmacokinetics (PK), and safety of two dose levels of CSJ117 in comparison to placebo. For this, the impact of CSJ117 on disease symptom burden and lung function will be explored.

DETAILED DESCRIPTION:
This is a randomized, participant- and investigator-blinded, placebo-controlled, parallel group, multicenter study with two fixed-dose levels of CSJ117 (4 mg, 8 mg) administered once-daily via oral inhalation over 12 weeks in participants with COPD, prone for exacerbations and symptomatic at baseline despite background maintenance triple therapy (inhaled corticosteroids/long acting beta-2 agonist/long acting muscarinic antagonist (ICS/LABA/LAMA) combination, standard of care in this population) for at least three months prior to screening.

The study will include:

* Screening period of up to 2 weeks to assess eligibility.
* Run-in period of 4 weeks where participants will be placed on fixed-dose triple background therapy (ICS/LABA/LAMA) that will be used until the patient's last study treatment.
* Treatment period of 12 weeks. Participants will be stratified by eosinophil levels and then randomized 1:1:1 to either 4 mg CSJ117, 8 mg CSJ117, or placebo.
* Follow-up period of 55 days following the last dose of study drug. The primary objective of the study is to assess the effect of CSJ117 on disease/symptom burden after 12 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male and female COPD patients aged ≥40 years, who have signed an Informed Consent Form prior to initiation of any study-related procedure
* Current or ex-smokers who have a smoking history of at least 10 pack years
* Patients who have been treated with a triple combination of LABA/LAMA/ICS for the last 3 months prior to screening
* Patients with a documented diagnosis of COPD for at least 1 year prior to screening visit

Exclusion Criteria:

* Patients with a past or current medical history of asthma
* Patients who have had a COPD exacerbation that required treatment with antibiotics and/or oral corticosteroids and/or hospitalization, or a respiratory tract infection in the 4 weeks prior to screening, or hospitalization between screening and prior to treatment.
* Use of other investigational drugs (approved or unapproved) within 30 days or 5 half-lives prior to screening, or until the expected pharmacodynamic effect has returned to baseline (e.g., biologics), whichever is longer; or longer if required by local regulations
* Pregnant or nursing (lactating) women, and women of childbearing potential not willing to use acceptable effective methods of contraception during study participation
* Patients with a body mass index (BMI) of more than 40 kg/m2 Other protocol-defined inclusion/exclusion criteria may apply

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2021-09-24 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline in E-RS score | Baseline, 12 weeks
  The Evaluating Respiratory Symptoms (E-RS) scale is based on the 11 respiratory symptom items included in the EXACT Tool (a validated 14-item electronic questionnaire). These 11 items generate a total score of 0-40, with higher scores indicating more severe respiratory symptoms.

SECONDARY OUTCOMES:
Change from baseline in CAT score | Baseline, 12 weeks
  The COPD assessment test (CAT) is a short instrument used to quantify the symptom burden of COPD and will be used to assess the health status of participants. The assessment consists of 8 items, each presented as a semantic 6-point differential scale, providing a total score out of 40. A higher score indicates a worse health status.
Change from baseline in SGRQ-C score | Baseline, 12 weeks
  The St. George Respiratory Questionnaire for COPD patients Specific Version (SGRQ-C) contains 40 items divided into two parts covering three aspects of health related to COPD: symptoms, activity and impacts. Total score ranges between 0 and 100, with higher scores indicating greater impairment of health status.
Response in E-RS in total score decrease from baseline | Baseline, 12 weeks
  To assess the number of patients who responded to treatment
Response in CAT in total score decrease from baseline | Baseline, 12 weeks
  To assess the number of patients who responded to treatment
Response in SGRQ-C in total score decrease from baseline | Baseline, 12 weeks
  To assess the number of patients who responded to treatment
Change from baseline in trough FEV1 after 2, 6, and 12 weeks of treatment | Baseline, 2, 6 and 12 weeks
  Forced expiratory volume in 1 second (FEV1) is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation, measured through spirometry testing.
Puffs of rescue medication per day | 12 weeks
  To assess use of rescue medication
Time to COPD exacerbations via EXACT | 12 weeks
  Time to COPD exacerbations based on EXACT.
Rate and severity of COPD exacerbations via EXACT | 12 weeks
  Rate and severity of COPD exacerbations based on the Exacerbations of chronic obstructive pulmonary disease tool (EXACT).
Time to COPD exacerbations via HCRU | 12 weeks
  Time to COPD exacerbations based on HCRU
Rate and severity of COPD exacerbations via HCRU | 12 weeks
  Rate and severity of COPD exacerbations based on the Health Care Resource Utilization (HCRU).
Pre-dose trough concentration (Ctrough) of CSJ117 | 12 weeks
  To assess pharmacokinetic (PK) parameters of CSJ117 based on total serum concentrations.
Accumulation ratio (Racc) of CSJ117 | 12 weeks
  To assess PK parameters of CSJ117 based on total serum concentrations.
Measuring anti-drug antibodies | 12 weeks
  To assess the immunogenicity of CSJ117

CONTACTS AND LOCATIONS:
Locations (15):
- United States (7):
  - Novartis Investigative Site, Andalusia, Alabama
  - Novartis Investigative Site, Crowley, Louisiana
  - Novartis Investigative Site, New Orleans, Louisiana
  - Novartis Investigative Site, Saint Charles, Missouri
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Huntersville, North Carolina
  - Novartis Investigative Site, Shelby, North Carolina
- Novartis Investigative Site, South Brisbane, Queensland, Australia
- Novartis Investigative Site, Sainte-Foy, Quebec, Canada
- Novartis Investigative Site, Ostrava Poruba, Czech Republic, Czechia
- Hungary (3):
  - Novartis Investigative Site, Balassagyarmat
  - Novartis Investigative Site, Gödöllő
  - Novartis Investigative Site, Szeged
- Japan (2):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Naka-gun, Ibaraki

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.